CLINICAL TRIAL: NCT04578171
Title: Type and Mechanisms of Residual Asthma Exacerbations in Patients Treated With Mepolizumab
Brief Title: Residual Exacerbations With Mepolizumab
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Andréanne Côté, Respirologist-intensivist, Laval University
Other Study IDs: CÉR21903
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: exacerbation; inflammation; monoclonal antibody
MeSH Terms: conditions — Asthma; Inflammation | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Subjects with severe asthma treated with mepolizumab
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — 100 mg subcutaneous injections every four weeks
  Other Names: nucala

SUMMARY:
This will be a two-year prospective study to characterize the nature of the remaining asthma exacerbations in patients treated with mepolizumab. Participants will be assessed every six months from pre- until two years of treatment in addition to whenever they experience an exacerbation of asthma during the study period. During these visits, various clinical, physiological and inflammatory outcomes will be assessed.

DETAILED DESCRIPTION:
Before initiation of mepolizumab, a recording of patient's demographics, clinical, physiological and inflammatory features will be recorded. All subjects will be reassessed for the above measures at 6, 12, 18 and 24 months.

In addition to the above visits, patients will be assessed every time they experience either moderate or severe exacerbation of asthma over the treatment period.

Based on the percentage of sputum eosinophils and neutrophils, the type of inflammatory exacerbation will be determined

ELIGIBILITY:
Inclusion Criteria:

* With a proven diagnosis of severe asthma as defined by the Canadian Thoracic Society
* Eligible for mepolizumab treatment
* Able and willing to sign the informed consent form

Exclusion Criteria:

* Any respiratory disease apart from asthma
* Confounding comorbidities sur as eosinophilic granulomatosis with polyangiitis (EGPA) or hypereosinophilic syndrome

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe asthma treated with mepolizumab at the IUCPQ-UL a tertiary care center from the Quebec city area.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eosinophilic vs non-eosinophilic remaining exacerbation during the treatment period | Between baseline and month 24
  Eosinophilic exacerbation defined as >=3% sputum eosinophils. Ratio of eosinophilic vs non eosinophilic asthma exacerbation

SECONDARY OUTCOMES:
Change from baseline in asthma control on the Asthma Control Questionnaire (ACQ-5) at 24 months | Baseline and month 24
  The ACQ-5 is a validated, self-reported questionnaire assessing asthma control over the last week. Possible scores range from 0 (complete control) to 5 (no control). Change = (Month 24 score - baseline score)
Change from baseline in post-bronchodilator forced expiratory volume in one second (FEV1) at 24 months | Baseline and month 24
  Value of FEV1 measured after inhalation of 400ug of salbutamol. Recorded in Li. (Month 24 FEV1 value - baseline FEV1 value)
Change from baseline in post-bronchodilator FEV1/forced vital capacity (FVC) ratio at 24 months | Baseline and month 24
  Value of FEV1/FVC measured after inhalation of 400 ug of salbutamol. (Month 24 value - baseline value)
Change from baseline in fraction of exhaled nitric oxide (FeNO) levels at 24 months | Baseline and month 24
  Recorded in ppb using the mean of two reproducible measurements. (Month 24 value - baseline value)
Change from baseline in percentage of sputum eosinophils at 24 months | Baseline and month 24
  Determined from induced sputum analysis. (Month 24 sputum eosinophil percentages - baseline sputum eosinophil percentages)
Change from baseline in percentage of sputum neutrophils | Baseline and month 24
  Determined from induced sputum analysis. (Month 24 sputum neutrophil percentages - baseline sputum neutrophil percentages).

CONTACTS AND LOCATIONS:
Overall Officials: Andréanne Côté, MD, Principal Investigator — IUCPQ-UL
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No